CLINICAL TRIAL: NCT05341479
Title: Department of Otorhinolaryngology, Eye & ENT Hospital
Brief Title: An Observational Study of Clinical Treatments for Patients With Oropharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, LeiTao, Director, Eye & ENT Hospital of Fudan University
Other Study IDs: FD-EENT-2022036
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Oropharynx Carcinoma
Keywords: Oropharynx carcinoma; Treatment; Survival outcomes
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Surgical Procedures, Operative; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Tumor tissue (If available), Para-tumor tissue (If available)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Surgical treatment for early-stage OPC: Early-stage OPC patients treated with surgery according to proper indications (CSCO 2021 and NCCN 2021).
  Interventions: Procedure: Surgery for early-stage OPC
- RT treatment for early-stage OPC: Early-stage OPC patients treated with radiotherapy (RT) according to proper indications (CSCO 2021 and NCCN 2021).
  Interventions: Radiation: RT for early-stage OPC
- CRT treatment for advanced OPC: Advanced OPC patients treated with chemoradiotherapy (CRT) according to proper indications (CSCO 2021 and NCCN 2021).
  Interventions: Radiation: CRT for advanced OPC
- Surgical treatment for advanced OPC: Advanced OPC patients treated with surgery according to proper indications (CSCO 2021 and NCCN 2021).
  Interventions: Other: Surgery for advanced OPC
- Neoadjuvant treatment for advanced OPC: Advanced OPC patients treated with neoadjuvant treatment according to proper indications (CSCO 2021 and NCCN 2021).
  Interventions: Procedure: Neoadjuvant treatment for advanced OPC

INTERVENTIONS:
Procedure: Surgery for early-stage OPC — The treatment strategy for patients should be discussed by the multidisciplinary team with the goal of maximizing survival with preservation of appearance and function and planned based on the tumor extension as ascertained by clinical evaluation and careful interpretation of appropriate imaging examinations.
  Early-stage OPC patients (T1-2,N0) enrolled in this group will be treated with surgical resection. The surgical techniques of the primary tumor include transoral robotic surgery, conventional transoral surgery, transoral laser microsurgery (e.g., CO2 laser resection), and open surgery. Ipsilateral neck dissection should be performed for patients enrolled in this group. For patients with OPC at or approaching the midline, bilateral neck dissection should be strongly considered.
  Postoperative radiotherapy (RT) or system therapy/RT should be considered for patients with adverse features (e.g., extranodal extension, perineural invasion or vascular invasion).
  Groups: Surgical treatment for early-stage OPC
Radiation: RT for early-stage OPC — The treatment strategy for patients should be discussed by the multidisciplinary team with the goal of maximizing survival with preservation of appearance and function and planned based on the tumor extension as ascertained by clinical evaluation and careful interpretation of appropriate imaging examinations.
  Early-stage OPC patients (T1-2,N0) enrolled in this group will be treated with RT.
  Groups: RT treatment for early-stage OPC
Radiation: CRT for advanced OPC — The treatment strategy for patients should be discussed by the multidisciplinary team with the goal of maximizing survival with preservation of appearance and function and planned based on the tumor extension as ascertained by clinical evaluation and careful interpretation of appropriate imaging examinations.
  Advanced OPC patients (T1-2,N1-3/T3-4,N0-3) enrolled in this group will be treated with CRT.
  Groups: CRT treatment for advanced OPC
Other: Surgery for advanced OPC — The treatment strategy for patients should be discussed by the multidisciplinary team with the goal of maximizing survival with preservation of appearance and function and planned based on the tumor extension as ascertained by clinical evaluation and careful interpretation of appropriate imaging examinations.
  Advanced OPC patients (T1-2,N1-3/T3-4,N0-3) enrolled in this group will be treated with surgical resection. The surgical techniques of the primary tumor include transoral robotic surgery, conventional transoral surgery, transoral laser microsurgery, and open surgery. Ipsilateral neck dissection should be performed for patients enrolled in this group. For patients with OPC at or approaching the midline, bilateral neck dissection should be strongly considered.
  Postoperative radiotherapy (RT) or system therapy/RT should be considered for patients with adverse features (e.g., pT3 or pT4 primary, pN2 or pN3 nodal disease, extranodal extension, or vascular invasion).
  Groups: Surgical treatment for advanced OPC
Procedure: Neoadjuvant treatment for advanced OPC — The treatment strategy for patients should be discussed by the multidisciplinary team with the goal of maximizing survival with preservation of appearance and function and planned based on the tumor extension as ascertained by clinical evaluation and careful interpretation of appropriate imaging examinations.
  Advanced OPC patients (T1-2,N1-3/T3-4,N0-3) enrolled in this group will be treated with neoadjuvant treatment. The subsequent treatments include RT, system therapy/RT, and surgical resection with or without postoperative adjuvant therapy.
  Groups: Neoadjuvant treatment for advanced OPC

SUMMARY:
This is a prospective, observational study evaluating the effect and efficiency of different clinical treatments for patients with oropharyngeal carcinoma (OPC). The selection of treatment for individual patient is based on tumor characteristics (tumor size and tumor location), a complete assessment of therapeutic effects (treatment effectiveness, possible dysfunction after operation, function maintenance, complications, etc.), and the preferences of doctors and patients.

DETAILED DESCRIPTION:
For early-stage oropharyngeal carcinoma (T1-2,N0), radiotherapy or resection of the primary tumor (transoral laser microsurgery, transoral robotic surgery, conventional transoral surgery, and open surgery) with ipsilateral or bilateral neck dissection are performed according to the guidelines of Chinese society of clinical oncology (CSCO, version 2021) and the NCCN guidelines (version 2021). Postoperative radiotherapy (RT) or chemoradiotherapy (CRT) should be considered for patients with adverse features (e.g., extranodal extension, positive margins, perineural invasion or vascular invasion).

For advanced oropharyngeal carcinoma (T1-2,N1-3/T3-4,N0-3), chemoradiotherapy (CRT), resection of the primary tumor (transoral robotic surgery, conventional transoral surgery, transoral laser microsurgery, and open surgery) with ipsilateral or bilateral neck dissection or neoadjuvant therapy with appropriate therapy (surgical resection, RT or CRT) are performed according to the CSCO guidelines (version 2021) and the NCCN guidelines (version 2021). Postoperative radiotherapy (RT) or chemoradiotherapy (CRT) should be considered for patients with adverse features (e.g., pT3 or pT4 primary, pN2 or pN3 nodal disease, extranodal extension, positive margins, perineural invasion or vascular invasion).

This study aims to evaluate and compare the clinical outcomes of different medical treatments in patients with same TNM stage disease, overall and stratified by HPV expression. Demographic and clinicopathological characteristics of patients enrolled were also collected to assess their associations with treatment strategies and prognoses. The rates of overall survival, disease specific survival, disease free survival, local control, regional control, and progress-free survival are analyzed in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Oropharyngeal cancer: Base of Tongue/Tonsil/Posterior Pharyngeal Wall/Soft Palate;
* T1, T2, T3, and T4 stage.
* Age 18 - 90.
* Male or female.
* Good compliance.
* No other severe related diseases that may impact the treatment (such as other tumors, severe heart, lung and central nervous system diseases, etc.).
* Negative pregnancy test (for female patients with fertility).
* Male patients with fertility and female patients with fertility and pregnancy risk must agree to use contraceptive methods throughout the study period, and continued until at least 6 months after the last dose of cisplatin. Female patients do not have fertility. Female patients with postmenopausal status.

Exclusion Criteria:

* Patients who have previously been diagnosed with immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related diseases.
* Patients with a known history of active tuberculosis (TB).
* Pregnant women or lactating women.
* The doctors believes that it is inappropriate for patients to participate in the trial: having, for example, severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including recent time [within the past year] or active suicidal ideation or behavior).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, observational study involves patients with T1-T4 stages oropharyngeal carcinoma, and we aim to evaluate and compare the oncological outcomes of different clinical treatments in patients with same TNM stage disease, overall and stratified by HPV expression. Demographic and clinicopathological characteristics of patients enrolled are also collected to assess their associations with treatment strategies and prognoses.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | Three years
  The time between the treatment and the date of death from any causes

SECONDARY OUTCOMES:
3-year local control survival | Three years
  The time between the treatment and the first evidence of local recurrence
3-year regional control | Three years
  The time between the treatment and the first evidence of regional recurrence
3-year disease specific survival | Three years
  The time between the treatment and the date of death from oropharyngeal cancer
3-year disease free survival | Three years
  The time between the treatment and the first evidence of disease recurrence, metastasis or death from any cause
3-year progress-free survival | Three years
  The time between the treatment and the date of first documented disease progression or death from any cause
Quality of Life post treatment | One year and three years post treatment
  Quality of life as assessed with the MD Anderson Dysphagia Inventory (MDADI)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Tao, Dr., Study Chair — Department of Otorhinolaryngology, Eye & ENT Hospital, Fudan University, Shanghai, China
Locations (1):
- Department of Otorhinolaryngology, Eye & ENT Hospital, Shanghai, Shanghai Municipality, China